CLINICAL TRIAL: NCT04425187
Title: Bevacizumab Combined With Gefitinib in the Treatment of Advanced NSCLC Clinical Study of L858R Positive Mutation Patients
Brief Title: Bevacizumab Combined With Gefitinib in the Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEVA-FLFX-001
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: PFS
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gefitinib (Active Comparator)
  Interventions: Drug: Gefitinib
- gefitinib&bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab Combined With Gefitinib

INTERVENTIONS:
Drug: Gefitinib — gefitinib 250mg (1 tablet), once a day，PO
  Arms: gefitinib
Drug: Bevacizumab Combined With Gefitinib — Bevacizumab Combined With Gefitinib
  Arms: gefitinib&bevacizumab

SUMMARY:
To compare the efficacy and safety of gefitinib combined with bevacizumab and gefitinib in the treatment of L858R positive mutation in exon 21 of EGFR gene in advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender unlimited.
2. NSCLC was confirmed by histology or cytology, and it was evaluated as stage IIIB-IV local advanced, recurrent or metastatic patients who could not be treated surgically. Note: ① the diagnosis result of NSCLC based on sputum cytology needs to be confirmed by immunohistochemistry; ② the current disease should be treated by radiotherapy as the first choice The subjects whose treatment strategy or follow-up target focus judged by the researchers should take radiotherapy as the first treatment strategy should not be selected.
3. No systemic anti-tumor therapy was received for locally advanced, recurrent or metastatic NSCLC.
4. According to the method of second-generation sequencing, L858R point mutation in exon 21 of EGFR gene was found in primary NSCLC with or without any other coexisting mutations.
5. Within 28 days before randomization, at least one measurable lesion was selected according to the RECIST v1.1 standard (see Appendix 1); for the lesions that had previously received radiotherapy, only when there was clear disease progression 3 months after the end of radiotherapy, can they be selected as target lesions.
6. ECoG general condition score is 0-1 (see Appendix 2).
7. Expected survival ≥ 12 weeks.
8. Patients receiving radiotherapy can be included in the group if they meet the following conditions:

   There was no history of lung disease radiotherapy within 28 days before randomization; L. for radiotherapy outside the chest area, the interval from the end of final radiotherapy to at least 28 days before randomization, and all toxic reactions have recovered.
9. Good blood function within 14 days before randomization:

L. the absolute neutrophil count (ANC) was ≥ 1.5 × 109 / L (without the support of granulocyte colony stimulating factor) and; L lymphocyte count ≥ 0.5 × 109 / L and; 1. Platelet count ≥ 100 × 109 / L and; Hemoglobin ≥ 9 g / dl (in order to reach this standard, patients can receive blood transfusion).

10. Good liver function within 14 days before randomization: L) total bilirubin ≤ 1.5 × upper normal limit (ULN) and;

1. Ast, ALT and ALP of patients without liver metastasis were less than 2.5 × ULN; ast, ALT and ALP of patients with liver metastasis were less than 5 × ULN.

11. Good renal function within 14 days before randomization:

1. Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 45 ml / min and; The urine test paper of urine protein was less than 2 +. If the baseline urine analysis of proteinuria patients is ≥ 2 +, 24-hour urine sample collection must be completed, and 24-hour urine protein ≤ 1 g; serum albumin ≥ 25 g / L.

12. Within 14 days before randomization, INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN. 13. Heart function meets the requirement of left ventricular ejection fraction (LVEF) ≥ 50%.

14. Fertile women: during the treatment period and within 6 months after the last administration, they agreed to abstinence (no heterosexual sexual intercourse) or use contraceptive methods (contraceptive methods with a failure rate of less than 1%). If a postmenopausal woman has not reached the postmenopausal state (menopausal time ≥ 12 months, no other reason except menopause) and has not undergone sterilization (removal of ovaries and / or uterus), she is defined as a woman with fertility.

15. Male: for male patients with fertility of female partners or pregnancy of female partners, they agree to abstinence (no heterosexual sexual intercourse) or use condoms within 6 months after the last administration, and agree not to donate sperm.

16. Sign the informed consent voluntarily. 17. The researchers judged that they could comply with the research plan.

-

Exclusion Criteria:

1. Histology or cytology confirmed mixed adenocarcinoma with squamous cells as the main component (the proportion of squamous cells ≥ 10%).
2. There was a history of malignancy (except NSCLC) in the first 5 years before randomization, except for malignancies with negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as cervical carcinoma in situ, non melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ or stage I uterine cancer, which were treated appropriately.
3. Previous hypertensive crisis, hypertensive encephalopathy, or uncontrolled hypertension (blood pressure: systolic pressure > 150 mmHg and / or diastolic pressure > 100 mmHg).
4. The tumor invades the main blood vessels. Researchers or local radiologists must rule out evidence that the tumor is completely adjacent to, surrounding, or extending into the lumen of a major artery, such as the pulmonary artery or superior vena cava.
5. Any other disease, neurological or metabolic dysfunction; medical examination or laboratory finding that a disease or condition is suspected, which prohibits the use of the test drug or exposes the patient to a high risk of treatment-related complications.
6. It is highly suspected that there are patients with idiopathic pulmonary fibrosis, organic pneumonia, drug-related pneumonia, idiopathic pneumonia, active pneumonia or active tuberculosis.
7. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently) allows patients to retain catheters.
8. History of hereditary bleeding constitution or coagulation disorder or other evidence of increased bleeding risk.
9. There are non healing wounds, active ulcers or fractures.
10. Patients with tracheoesophageal fistula, gastrointestinal perforation or gastrointestinal fistula, and intraperitoneal abscess in the first 6 months were randomly assigned.
11. Cardiovascular diseases with clinical significance (such as active), including but not limited to TIA (within 6 months before screening), myocardial infarction (within 6 months before screening), unstable angina, congestive heart failure with New York Heart Association classification ≥ level II (see Appendix 3), and serious arrhythmias beyond the control of drugs.
12. Within 3 months before randomization, there was a history of hemoptysis ≥ 2 levels, that is, the blood volume of each bleeding event was > 2.5ml.
13. Evidence of central nervous system metastasis, except for patients without any symptoms or patients with symptoms but stable condition, at least 28 days after treatment of central nervous system metastasis.
14. Major surgery (including open biopsy) or severe trauma was performed within 28 days prior to randomization, or was expected to be performed during study treatment.

Severe infections occurring within 28 days prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.

16 aspirin (325 mg / day) or other non steroidal anti-inflammatory drugs known to inhibit platelet function are currently or recently used (within 10 days before bevacizumab was first used).

17 full dose oral or parenteral anticoagulants or thrombolytic agents are currently or recently used (within 10 days prior to the first use of bevacizumab). Preventive use of anticoagulants is permitted.

18. Core biopsies or other minor operations were performed within 7 days prior to randomization, but vascular access devices were not included. Vascular access devices should be placed at least 2 days before the start of study treatment.

19. Those who are known to be allergic to bevacizumab, gefitinib and their excipients, or to Chinese hamster ovarian cell products or other recombinant human or humanized antibodies.

20. Those who were confirmed to be HCV positive, HIV positive, syphilis positive, or HBsAg positive during the screening period, and whose HBV DNA titer in the peripheral blood was ≥ 1000 copies / L.

21. Pregnancy or lactation, or pregnancy planning during the study. 22. Those who participated in any other clinical trial and took the trial drug treatment within 30 days before randomization.

23. The investigator determined that the risk of the subject was greater than any other benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  The PFS of gefitinib combined with bevacizumab and gefitinib alone were compared in patients with L858R mutation in exon 21 of EGFR gene in stage IIIB-IV local advanced, recurrent or metastatic NSCLC.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhao X, Wu X, Wang H, Yu H, Sun S, Hu Z, Lin Y, Zhang Y, Yu B, Wu Z, Xiong K, Liu C, Wang S, Bao H, Ou Q, Wang J. Evaluation of gefitinib alone or combined with bevacizumab in patients with EGFR L858R-positive advanced non-squamous non-small cell lung cancer: an open-label, randomized, phase 2 trial (BEVA-FLFX-001) with exploratory analysis of plasma biomarkers. Transl Lung Cancer Res. 2025 Oct 31;14(10):4315-4330. doi: 10.21037/tlcr-2025-545. Epub 2025 Oct 29. PMID 41234598